CLINICAL TRIAL: NCT05379348
Title: Davos Alzheimer's Collaborative Study: Sequential Administration of Digital Testing To Screen For Cognitive Impairment Followed By Blood Based Biomarkers To Assist With Timely Detection And Accurate Diagnosis Of Alzheimer's Disease
Acronym: DAC
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Davos Alzheimer's Collaborative (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1811673
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General study participants (patients)
  Interventions: Other: Cognitive Assessment
- Healthcare Practitioners
- Pre-Program Chart Audits (100 patients what will be chart audited)

INTERVENTIONS:
Other: Cognitive Assessment — Montreal Cognitive Assessment - MoCA, which is a cognitive screening tool that assesses: memory, concentration, language, and orientation to time and place. this written cognitive test should take no more than 20 minutes.
  Other Names: MoCA
  Groups: General study participants (patients)

SUMMARY:
The purpose of this study is to investigate how we can detect Alzheimer's disease early by using an online memory test and a simple blood test. These new methods for early diagnosis could allow people to begin treatment sooner, with the potential to improve the lives of millions of people.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet the following criteria for entry into the study:

1. Male or female > 65 years of age at the time of consent;
2. Understand and voluntarily sign an informed consent form;

Inclusion criteria is assessed at both e-consent (assessed by participant's self-reporting of age and understanding) and in-person consent at TRI (assessed by clinical research coordinators in TRI).

Exclusion Criteria

Subjects who meet any of the following criteria will not be eligible for entry into the study:

1. Subjects who are unable to hear and see well enough to complete the assessments;
2. Prior diagnosis of dementia or Alzheimer's disease documented in their medical record and/or as diagnosed by a physician; Exclusion criteria is assessed by by participant's self-reporting of understanding and not having a prior diagnosis of dementia at the time of e-consentand visit 1 at TRI. ).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy male and females ages >65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1423 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quantify the proportion of individuals at least 65 years old with cognitive impairment | Less than 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Smith, MD, Principal Investigator — Study PI
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

REFERENCES:
- See also: Related Info — https://www.adventhealthresearchinstitute.com/research/translational-research